CLINICAL TRIAL: NCT01829321
Title: Exploratory, Phase II, Randomized, Double-blind, Placebo-controlled, Proof-of-Concept Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics and Pharmacodynamics of GLPG0974 in Subjects With Mild to Moderate Ulcerative Colitis
Brief Title: Safety, Efficacy, Pharmacokinetic and Pharmacodynamic Study of GLPG0974 in Subjects With Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG0974-CL-201; 2012-005521-73 (EudraCT Number)
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — 4-(((R)-1-(benzo(b)thiophene-3-carbonyl)-2-methyl-azetidine-2-carbonyl)-(3-chloro-benzyl)-amino)-butyric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLPG0974 (Experimental): 1 capsule of 200 mg GLPG0974 twice daily
  Interventions: Drug: GLPG0974
- Placebo (Placebo Comparator): 1 capsule placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG0974 — 1 capsule in the morning and 1 capsule in the evening with food during 28 days
  Arms: GLPG0974
Drug: Placebo — 1 capsule in the morning and 1 capsule in the evening with food during 28 days
  Arms: Placebo

SUMMARY:
* Approximately 45 patients suffering from mild to moderate ulcerative colitis will be examined for any side effects (safety and tolerability) that may occur when taking GLPG0974 or matching placebo (2:1 ratio) for 28 days.
* During the course of the study, patients will also be evaluated for improvement of disease activity by different efficacy measures, the amount of GLPG0974 present in the blood determined (PK) and the effects of GLPG0974 on selected biomarkers (PD) in the blood, colon biopsies and faeces will be explored.

ELIGIBILITY:
Key Inclusion Criteria:

* Men or women between 18 to 75 years of age inclusive, on the day of signing the informed consent with a documented history of UC.
* Presence of mild-to-moderately active ulcerative colitis as evidenced by clinical signs and endoscopy.
* Medication: 5-ASA.
* Absence of infectious colitis.

Key Exclusion Criteria:

* History of sensitivity to any component of the study drug
* Any concurrent illness, condition, disability or clinically significant abnormality (including lab tests) that represents a safety risk , may affect the interpretation of data, or may prevent the subject to safely complete the assessments
* Positive serology for HIV 1 or 2 or hepatitis B or C, or any history of HIV or hepatitis.
* History of active infections requiring intravenous antibiotics within the past four weeks prior to randomization.
* History of bowel surgery, or presence or history of intestinal malignancy.
* Suspicion of Crohn's disease, indeterminate colitis, microscopic colitis, ischaemic colitis or radiation-induced colitis.
* History of lower GI bleeding disorder, other than UC.
* A history of significant psychological, neurologic, hepatic, renal, endocrine, cardiovascular, gastrointestinal (other than UC), pulmonary or metabolic disease.
* History of tuberculosis (TB) infection.
* Treatment with systemic corticosteroids within 1 week prior to randomization.
* Treatment with TNF-α inhibitors or other biologics within 2 months prior to randomization.
* Treatment with immunosuppressants, initiated or changed within 3 months prior to randomization .
* Current use of probiotic or prebiotic preparations
* Regular daily use of NSAIDs, within 7 days prior to randomization.
* Administration of any experimental therapy within 90 days or 5x the half-life.
* History of drug or alcohol abuse.
* Pregnant or lactating women.
* Medical, psychiatric, cognitive, or other conditions that compromise the subject's ability to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Screening up to Follow up (14 days after last dosing)
  To evaluate the safety and tolerability of GLPG0974 in terms of the number of adverse events reported
Changes in physical exam measures | Screening up to Follow up (14 days after last dosing)
  To evaluate the safety and tolerability of GLPG0974 in terms of the changes in physical exam measures reported
Changes in vital signs as measured by heart rate, blood pressure and oral temperature | Screening up to Follow up (14 days after last dosing)
  To evaluate the safety and tolerability of GLPG0974 in terms of the changes in vital signs as measured by heart rate, blood pressure and oral temperature reported
Changes in 12-lead ECG measures | Screening up to Follow up (14 days after last dosing)
  To evaluate the safety and tolerability of GLPG0974 in terms of the changes in 12-lead ECG measures reported
Changes in blood safety lab parameters | Screening up to Follow up (14 days after last dosing)
  To evaluate the safety and tolerability of GLPG0974 in terms of changes in blood safety lab parameters reported
Changes in urine safety lab parameters | Screening up to Follow up (14 days after last dosing)
  To evaluate the safety and tolerability of GLPG0974 in terms of changes in urine safety lab parameters reported

SECONDARY OUTCOMES:
Changes in (partial) Mayo clinical disease activity score | From Day 1 to Day 29
  To evaluate the efficacy of GLPG0974 in terms of changes in (partial) Mayo clinical disease activity score reported
Changes in histopathological clinical activity score in colon biopsies | Day 1 and Day 29
  To evaluate the efficacy of GLPG0974 in terms of changes in histopathological clinical activity score (Geboes score) in colon biopsies reported
The amount of GLPG0974 in plasma over time after multiple oral doses of GLPG0974 | Day 8, Day 15 and Day 29
  To evaluate the amount of GLPG0974 in plasma over time after multiple oral doses of GLPG0974 - pharmacokinetics (PK) in ulcerative colitis patients
Changes in the levels of faecal calprotectin over time after multiple oral doses of GLPG0974 | Screening up to Day 29
  To evaluate the changes in the levels of calprotectin in faeces over time after multiple oral doses of GLPG0974 - pharmacodynamics (PD) in ulcerative colitis patients
Changes in the levels of C-reactive protein in serum over time after multiple oral doses of GLPG0974 | Screening up to Day 29
  To evaluate the changes in the levels of C-reactive protein in serum over time after multiple oral doses of GLPG0974 - pharmacodynamics (PD) in ulcerative colitis patients
Changes in the levels of myeloperoxidase (MPO) in colon biopsies over time after multiple oral doses of GLPG0974 | Day 1 and Day 29
  To evaluate the changes in the levels of MPO in colon biopsies over time after multiple oral doses of GLPG0974 - pharmacodynamics (PD) in ulcerative colitis patients
Changes in the levels of predominant microbiota in faeces over time after multiple oral doses of GLPG0974 | Day 1 and Day 29
  To evaluate the changes in the levels of predominant microbiota in faeces over time after multiple oral doses of GLPG0974 - pharmacodynamics (PD) in ulcerative colitis patients
Changes in the levels of predominant microbiota in colon biopsies over time after multiple oral doses of GLPG0974 | Day 1 and Day 29
  To evaluate the changes in the levels of predominant microbiota in colon biopsies over time after multiple oral doses of GLPG0974 - pharmacodynamics (PD) in ulcerative colitis patients

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV
Locations (16):
- Belgium (4):
  - Imelda, Bonheiden
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
- Czechia (7):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Fakulní nemocnice Olomouc, Olomouc
  - Homolka Hospitál, Prague
  - Nemocnice Slaný, Slaný
  - Krajská zdravotní a.s., Masarykova nemocnice v Ústí nad Labem T. Bati a.s., Ústí nad Labem
  - Krajská nemocnice Tomáše Bati - Zlin, Zlín
  - Nemocnice Znojmo, Znojmo
- Latvia (3):
  - Latvijas Jūras Medicīnas Centrs, Riga
  - Rīgas slimnīca Bikor Holim, Riga
  - SIA Gremošanas slimību centrs "Gastro", Riga
- Slovakia (2):
  - Univerzitná nemocnica Bratislava, Bratislava
  - Fakultná Nemocnica Nitra, Nitra